CLINICAL TRIAL: NCT03017950
Title: Phase I Clinical Trial to Evaluate the Pharmacokinetic Drug-drug Interaction of CKD-330 and D086 in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug-drug Interaction of CKD-330 and D086
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 170DDI16017
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part1 (A) (Experimental): Number of Subjects: 10
  Number of days for Period 1: 8
  Number of days for Period 2: 8
  Number of days for wash-out between period 1 and period 2: 14
  IPs for Period 1: CKD-330
  IPs for Period 2: CKD-330 + D086
  Interventions: Drug: CKD-330; Drug: CKD-330 + D086
- Part1 (B) (Experimental): Number of Subjects: 10
  Number of days for Period 1: 8
  Number of days for Period 2: 8
  Number of days for wash-out between period 1 and period 2: 14
  IPs for Period 1: CKD-330 + D086
  IPs for Period 2: CKD-330
  Interventions: Drug: CKD-330; Drug: CKD-330 + D086
- Part2 (A) (Experimental): Number of Subjects: 30
  Number of days for Period 1: 8
  Number of days for Period 2: 8
  Number of days for wash-out between period 1 and period 2: 14
  IPs for Period 1: D086
  IPs for Period 2: CKD-330 + D086
  Interventions: Drug: D086; Drug: CKD-330 + D086
- Part2 (B) (Experimental): Number of Subjects: 30
  Number of days for Period 1: 8
  Number of days for Period 2: 8
  Number of days for wash-out between period 1 and period 2: 14
  IPs for Period 1: CKD-330 + D086
  IPs for Period 2: D086
  Interventions: Drug: D086; Drug: CKD-330 + D086

INTERVENTIONS:
Drug: CKD-330
  Arms: Part1 (A); Part1 (B)
Drug: D086
  Arms: Part2 (A); Part2 (B)
Drug: CKD-330 + D086

SUMMARY:
The purpose of the study is examining and comparing the pharmacokinetic drug interaction and safety of both single administration and combination administration of CKD-330 and D086 to healthy male subjects

DETAILED DESCRIPTION:
An open-label, randomized, multiple-dose, 2-sequence, 2-period, 2-treatment, crossover study

Part1: Examining how D086 affects pharmacokinetics of CKD-330. Part2: Examining how CKD-330 affects pharmacokinetics of D086.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males age of between 19 - 45 on the day of screening.
2. Body mass index(BMI) between 18.0 - 29.0 kg/m^2 and weight ≥ 55kg (Body mass index (BMI) = weight (kg) / height (m)^2)
3. Subjects in good health as determined by physical exams and medical examinations. No congenital or chronic diseases and no abnormal signs determined by medical examinations.
4. Not abnormal or not clinically significant lab values.
5. Subjects who signed informed consent form with good understandings after explanations by investigators.

Exclusion Criteria:

1. No history or presence of clinically significant cardiac, respiratory, neurological, endocrine, metal and renal diseases and liver and kidney diseases.
2. Subjects showing angioedema as an adverse reaction to ACE inhibitors
3. Primary Hyperaldosteronism
4. History or family history of myopathy
5. Subjects with mental diseases or drug addiction
6. Allergic reactions to candesartan or amlodipine or atorvastatin
7. Genetic problems in galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.
8. Hypotension(SBP ≤100mmHg or DBP≤55mnHg) or hypertension ( SNP ≥ 150mmHg, DBP ≥95mmHg) on the day of screening
9. Subjects who experienced gastrointestinal diseases or surgeries which can affect absorption of Investigational product
10. Subjects with abnormal lab values at least one below

    (AST or ALT>2 fold of upper normal limit, Total bilirubin>2 fold of upper normal limit, CPK>2 fold of upper normal limit, K <3.5mEq/L or >5.5mEq/L, Estimated Glomerular filtration rate<60mL/min/1.73m2 by Modification)
11. Continuous drinking (over 21 units/week, 1 unit= 10g=12.5mL of pure alcohol), heavy smoker(> 10 cigarettes per day) and unable to stop drinking during clinical trials
12. Subjects who previously participated in other clinical trials within 90 days
13. Subjects who donated whole blood within 60 days or donated component blood within 30 days or received blood transfusion within 30 days
14. Subjects who were administered below medications within 30 days (cyclosporin, erythromycin, clarithromycin, lopinavir, ritonavir, itraconazole, ketoconazole, rifampicin, barbiturate : theses medicines could affect absorption, metabolism, distribution and excretion of candesartan,amlodipine and atorvastatin)
15. Subjects who took any prescribed medications or oriental medicines within 14 days, or took any pharmacy medicines within 7 days.
16. Subjects who have taken any diets affecting absorption, metabolism, distribution and excretion of investigational products (especially grapefruit juice).
17. Subjects who are in conditions impossible participating in the clinical trials following other laboratory tests.
18. Unable to use contraceptions.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of Candesartan and Amlodipine | Day6, Day7, Day8, Day9, Day22, Day27, Day28, Day29 and Day30
AUCτ,ss of atorvastatin and 2-hydroxy atorvastatin | Day6, Day7, Day8, Day9, Day22, Day27, Day28, Day29 and Day30

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No